CLINICAL TRIAL: NCT05243589
Title: Effects of Proprioceptive Training in Addition to Routine Physical Therapy on Balance and Quality of Life in Patients With Diabetic Peripheral Neuropathy: a Randomized Controlled Trial
Brief Title: Effects of Proprioceptive Training in Addition to Routine Physical Therapy on Balance and Quality of Life in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Momna Asghar (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Sponsor-Investigator, Momna Asghar, Doctor, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/823/2021
Record Dates: First submitted 2022-02-05; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Neuropathy
Keywords: Neuropathy; Proprioceptive training; Balance; Quality of life; Physical therapy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A/ routine physical therapy and proprioceptive training (Experimental): Routine physical therapy and proprioceptive training is performed
  Interventions: Other: Proprioceptive training; Other: routine physical therapy
- Group B/ routine physical therapy (Active Comparator): Routine physical therapy
  Interventions: Other: routine physical therapy

INTERVENTIONS:
Other: Proprioceptive training — Proprioceptive training included exercises on different floor textures composed of 10 stations of exercises with the objective of stimulating the sole of the foot where participants had to coordinate gait by stepping with alternate feet on markers placed on the ground and the progression was manipulated through modifications of speed and direction.
  Sequence of materials was 10 cm-thick foam, wood box with beans, two-cm thick mat with a density lower than the foam, wood box with cotton, two-cm thick mat volunteers sat on a bench and trained feet flexors by grasping with the toes a towel put on the floor, Two proprioception balls was used with an eight cm diameter with external projections resting on the floor a box with grains and sandpaper. After that joint Positional Sense Exercises were performed.
  Arms: group A/ routine physical therapy and proprioceptive training
Other: routine physical therapy — Routine physical therapy included range of motion exercises for bilateral ankle joints (5 min.), functional balance training (15 min.) involving sit to stand (5 times); standing weight shift (5 times each); functional reach- sideway and anterior for touching targets set by the therapist (5 times each); bipedal heel rise for 20 seconds (5 times); unipedal standing for 15 seconds (5 times each) and unipedal standing with knee bending for 15 second (5 times each). Other exercises was practiced as wobble board training (6 min).

SUMMARY:
Objective of the study is to find out the effects of Proprioceptive training in addition to routine physical therapy on balance and quality of life in patients with Diabetic neuropathy.

Alternate Hypothesis:

There will be significant difference in effects of Proprioceptive training in addition to routine physical therapy on balance and Quality of life in patients with Diabetic neuropathy.

DETAILED DESCRIPTION:
It was a parallel designed single blinded randomized controlled trial conducted in the Green Poly Clinic Bahria town, Lahore, Pakistan using non probability convenient sampling. patients who met eligibility criteria was informed about the aim of study. consent form were signed by all participants.After baseline assessment ,participants were randomly assigned in two groups.(ratio 1:1) The calcualted sample size was 27 in each group. i.e. 54 ( 27 in each group). After adding 20% drop out the final size will become, 64( 32 in each group) using 95% level of significance and 80% power of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre-diagnosed DM for seven years.
* Male and female patients with type 2 diabetes.
* Patients with ≥2 DPN symptoms.
* Patients scored>2/13 on MNSI questionnaire.

Exclusion Criteria:

* Participants with Foot ulcers, Orthopedic or surgical problem in a lower limb, other neurological impairment and Major vascular complication,
* Severe vestibular dysfunction
* Participants with Severe retinopathy and Severe nephropathy,
* Inability to walk independently with or without an assistive device,
* Receiving any structured supervised physiotherapy intervention.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (assessing change in ability to balance at baseline, 4th week and at 6th week. | It was checked before the intervention started (after recruitment of patient) and then checked at the 4th week and then at the end of 6th weeks.
  It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4.0 denotes inability to complete the item, and 4 the ability to accomplish the task independently (total score range, 0-56; higher = better performance). Scores of less than 45 out of 56 are accepted as indicative of balance disorders in the elderly.
WHO Quality of Life Scale (WHOQOL BREF)( assessing change in quality of life at baseline, 4th and 6th week of intervention. | It was checked before the intervention started (after recruitment of patient) and then checked at the 4th week and then at the end of 6th weeks.
  The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centers, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally.It contains a total of 26 questions. To provide a broad and comprehensive assessment, one item from each of 24 facets contained in the WHOQOL-100 has been included.

CONTACTS AND LOCATIONS:
Overall Officials: Momna Asghar, MSPTN, Principal Investigator — University of Lahore
Locations (1):
- Atofa Rasheed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided